CLINICAL TRIAL: NCT03421275
Title: Intranasal Fentanyl and Esketamine for Treatment of Acute Pain in Minor Trauma Patients
Brief Title: Intranasal Esketamine and Fentanyl for Pain in Minor Trauma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anna Meuronen, MD (Other)
Responsible Party: Sponsor-Investigator, Anna Meuronen, MD, Principal Investigator, Hospital District of Helsinki and Uusimaa
Organization: Hospital District of Helsinki and Uusimaa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FK_0001
Record Dates: First submitted 2018-01-18; First posted 2018-02-05 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Acute Pain Due to Trauma
Keywords: fentanyl; esketamine; ketamine; analgesia; acute pain; minor trauma
MeSH Terms: conditions — Agnosia; Acute Pain | interventions — Esketamine; Fentanyl; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Esketamine (Experimental): intravenous anaesthetic and analgetic
  Interventions: Drug: Esketamine
- Fentanyl Citrate (Active Comparator): intravenous opioid analgetic
  Interventions: Drug: Fentanyl Citrate
- Saline Nasal (Placebo Comparator): intravenous "Natriumklorid b. Braun 9 mg/ml"
  Interventions: Drug: Saline Nasal

INTERVENTIONS:
Drug: Esketamine — anesthetic used as analgetic in subanesthetic doses given intranasally
  Other Names: Ketanest-S
  Arms: Esketamine
Drug: Fentanyl Citrate — intravenous fentanyl given intranasally
  Other Names: Fentanyl-Hameln
  Arms: Fentanyl Citrate
Drug: Saline Nasal — intravenous saline given intranasally as placebo
  Other Names: Natriumklorid b. Braun 9 mg/ml
  Arms: Saline Nasal

SUMMARY:
Intranasal esketamine, fentanyl and placebo are compared in treatment of acute pain in adult patients with minor trauma. Study is blinded randomized placebo-controlled parallel design.

ELIGIBILITY:
Inclusion Criteria:

* NRS 5 or more, minor trauma, no need for immediate iv cannulation, weight 45-115 kg

Exclusion Criteria:

* pregnancy, breastfeeding, head trauma, severe chronic obstructive pulmonary disease (COPD), gfr under 30, liver cirrhosis, mental illness other than mild/moderate depression, sleep apnea, unstable coronary artery disease (CAD), unstable heart failure (HF), intoxication, untreated hypertension, dementia, do not understand Finnish, contraindication to nasal spray, allergy to any of the medications, bradycardia, desaturation, suspected high intracranial pressure (ICP)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) change | 15 minutes and 30 minutes
  Numeric rating scale is used to measure pain intensity. Scale is from 0-10. 0 = no pain, 10 = worst imegeable

SECONDARY OUTCOMES:
Amount of patients with NRS change more than -2 | 15 min, 30 min, 60 min
  Amount of patients with NRS dropping more than 2 at time poin 15 minutes, 20 minutes and 60 minutes
Patient satisfaction (pain management) | 120 min
  Whole experience of pain management on NRS scale from 0-10 (0 = absolutely terrible, 10 = best imagenable)
Side effects | 120 min
Amount of study drug consumed (doses) | 120 min
  Amount of sturdy drug consumed as doses in the end of study period. One dose is determined by patient weight.
Need for rescue medication mg (oxycodone) | 120 min
  Amount of oral or intramuscular oxycodone consumption in the end of study period as milligrams

CONTACTS AND LOCATIONS:
Overall Officials: Anna Meuronen, MD,PhD, Principal Investigator — consultant
Locations (1):
- Hyvinkää Hospital, Hyvinkää, Finland

IPD SHARING:
Plan to Share IPD: No